CLINICAL TRIAL: NCT02012829
Title: Brief Intervention to Improve Colorectal Cancer Screening
Brief Title: Influence of a Brief Intervention on CRC Screening
Acronym: Hem-FMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Paris 7 - Denis Diderot (Other)
Responsible Party: Principal Investigator, Isabelle AUGER, Professor, University Paris 7 - Denis Diderot
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011/19NI
Record Dates: First submitted 2013-03-08; First posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer
Keywords: cancer, CRC screening, communication
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): GPs from practices in the control group are asked to continue their usual care, as if they were not participating in this trial. They had to send their patients list to the research team to calculate their eligible population. They were also asked to list all the gaiac Fecal occult blood test ( gFOBT) delivered during the six months period of the study.
- intervention (Active Comparator): GPs communication skills and CRC screening :the intervention was a four hours educational training for GPs of the intervention group focused on communication skills with a patients' centered care approach to improve patients participation at CRC screening
  Interventions: Behavioral: GPs communication skills and CRC screening

INTERVENTIONS:
Behavioral: GPs communication skills and CRC screening — GPs of the intervention group received a four hours educational training focused on patients' centered care to improve GPs communication skills and enhance patients'participation in CRC mass screening . Triangulation of all qualitative data was performed in order to develop educational material and training based on the six components of the Patient-Centered Clinical Method . Two different scenarios were developed: one for a compliant patient, another for a non-compliant patient. Two videos were made with doctor and simulated patient. Interactive methods were used to elaborate educational training including role playing, the presentation of the video followed by an interactive discussion.
  Arms: intervention

SUMMARY:
Qualitative data were collected from 5 General Practionners (GPs) focus groups, 24 patient interviews and 35 recorded consultations from 9 GPs to explore colorectal cancer (CRC) screening in France The qualitative data indicated that improvement was needed in patient-centered communication. Educational material was developed based on these triangulated data with two different scenarios to improve communication with patients: one for a compliant patient, another for a non compliant patient The hypothesis is that a brief intervention on GPs can improve the patients' participation rate to colorectal screening

Method : cluster randomized control trial (cluster unit : GPs practices) With a brief intervention on a randomized population of GPs in the district of Val d'Oise Inclusion criteria: GPs with a practice in the district of Val d'Oise and active in the colorectal mass screening

DETAILED DESCRIPTION:
a cluster randomized controlled parallel groups study was conducted in the Val d'Oise department in France All practices of the Val d'Oise department were eligible to participate. Among 585 practices, an independent biostatistician randomized 50 practices per arm in October 2011 according to a computer generated randomization list.Two team members phone called all the GPS of the randomized practices.

GPs from practices in the control group are asked to continue their usual care, as if they were not participating in this trial. GPs of both groups had to send their patients list to the research team to calculate their eligible population. They were also asked to list all the gFOBT delivered during the six months period of the study.

GPs of the intervention group received a four hours educational training focused on patients' centered care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion of GPs practices: All GPs practices of the Val d'Oise department in France were eligible to participate GPs using complementary therapies occasionally were allowed to participate

Exclusion Criteria:

Exclusion of GPs practices : practices were excluded when doctors used exclusively complementary therapies (acupuncture therapy, homeopathy….)

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
participation rate of patients for CRC screening | 7 months
  Comparison of the participation rate for patients for CRC screening among GPs belonging to the intervention group versus the participation rate for patients for CRC screening among GPs belonging to the control group

SECONDARY OUTCOMES:
GPs with a participation rate over 65% | 7 months
  the number of GPs who reached a patients participation rate of 65% during the study period because of the desirable level of uptake rate over 65% defined by the European guidelines of quality assurance in colorectal cancer screening
GPs participation rate over 45% | 7 months
  The number of Gps who reached a participation rate of 45% because of the acceptable level of uptake defined by the same guidelines , the number of gFOBT delivered by GPs during study period,

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AUGER, Professor, Principal Investigator — University Paris Diderot
Locations (1):
- University Paris Diderot, Paris, France